CLINICAL TRIAL: NCT07400653
Title: EVALUATING THE EFFICACY AND SAFETY OF MET097, A FULLY-BIASED ULTRA LONG-ACTING GLP-1RA, IN PEOPLE WITH OVERWEIGHT OR OBESITY AND TYPE 2 DIABETES: A PHASE 3, MULTI-CENTER RANDOMIZED PLACEBO-CONTROLLED TRIAL (VESPER-5)
Brief Title: A Study to Learn About the Study Medicine (PF-08653944) in People With Obesity or Overweight and Type 2 Diabetes (T2D)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C6491008; VESPER-5 (Other: Alias Study Number); 2025-523975-48-00 (Registry Identifier: CTIS (EU)); MET097-25-302 (Other: Alias Study Number); VESPER-5 (MET097-25-302) (Other: Alias Study Number)
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Overweight and/or Obesity; Overweight; Diabetes, Type 2; Type 2 Diabetes
Keywords: Overnutrition; Nutrition Disorders; Nutritional and Metabolic Diseases; Body Weight; Signs and Symptoms; Pathological Conditions, Signs and Symptoms; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Overweight; Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2; Overnutrition; Nutrition Disorders; Nutritional and Metabolic Diseases; Body Weight; Signs and Symptoms; Pathological Conditions, Signs and Symptoms; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment Arm 1 (Experimental): Participants will receive PF-08653944 by Subcutaneous Injection.
  Interventions: Drug: PF-08653944
- Treatment Arm 2 (Experimental): Participants will receive PF-08653944 by Subcutaneous Injection.
  Interventions: Drug: PF-08653944
- Treatment Arm 3 (Experimental): Participants will receive PF-08653944 by Subcutaneous Injection.
  Interventions: Drug: PF-08653944
- Placebo (Placebo Comparator): Participants will receive matching placebo by Subcutaneous Injection.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-08653944 — By Subcutaneous Injection
  Other Names: MET097
  Arms: Treatment Arm 1; Treatment Arm 2; Treatment Arm 3
Other: Placebo — By Subcutaneous Injection
  Arms: Placebo

SUMMARY:
The purpose of this clinical study is to learn about the safety and effects of the study medicine to help adults with obesity or overweight and type 2 diabetes lose weight. Being overweight or obese means carrying too much body weight. Type 2 diabetes is a condition where there is too much sugar in the blood.

The study medicine is given by a shot under the skin in the belly area. The participants will be trained to do this at home once every week.

About 660 out of 1000 adults will also receive the study medicine and about 330 out of 1000 adults will receive placebo. A placebo does not have any medicine in it but looks just like the medicine being studied. We will compare the experiences of people receiving the study medicine to those of the people who do not. This will help us assess if the study medicine is safe and effective.

People will take part in this study for about 21 months. During this time, they will have about 14 study visits at the site and 5 over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form (ICF)
* Male or female adults, aged ≥18 years
* Have a BMI at Screening of ≥27.0 kg/m2
* Have T2DM for at least 6 months before Screening based on participant reported history or documentation of the disease diagnostic criteria
* Have HbA1c value between ≥6.5% (48 mmol/mol) and ≤10.0% (86.0 mmol/mol) at Screening with stable therapy for at least 90 days prior to Screening/Visit 1. T2DM may be treated with:

  --Diet and exercise alone or in combination with: Any oral antidiabetic therapy per local labeling EXCEPT DPP-4 inhibitors. Participant may NOT be on GLP-1 agonists or insulin
* Participants must be motivated and willing to:

  * Self-inject study medication (or be aided by caregiver if needed),
  * Perform finger-stick glucose monitoring as required.
* Have a history of at least 1 self-reported unsuccessful dietary effort to lose body weight.

Exclusion Criteria:

* Female who is breastfeeding, or who is pregnant
* Unwilling or unable to follow contraceptive requirements
* Diagnosis of Type 1 diabetes, or any other types of diabetes except T2DM.
* Severe hypoglycemia and/or hypoglycemia unawareness within the 6 months prior to Screening
* Poorly controlled hypertension
* Have a prior or planned surgical treatment for obesity (excluding liposuction or abdominoplasty if performed >1 year prior to screening)
* Have taken within 3 months prior to randomization, medications (prescribed or over-the counter) intended to promote weight loss
* Are receiving or have received within 3 months prior to screening chronic (>2 weeks or 14 days) systemic glucocorticoid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 999 (Estimated)
Dates: Start 2026-02-12 (Estimated); Primary Completion 2027-10-12 (Estimated); Study Completion 2028-05-16 (Estimated)

PRIMARY OUTCOMES:
Percent Change from baseline in body weight | Baseline, Week 64

SECONDARY OUTCOMES:
Change from baseline in body weight | Baseline, Week 64 and 84
Change in HbA1c (%) from baseline | Baseline, Week 64 and 84
Percentage of Participants achieving ≥5% of body weight reduction from baseline | Baseline, Week 64 and 84
Percentage of Participants achieving ≥10% of body weight reduction from baseline | Baseline, Week 64 and 84
Percentage of Participants achieving ≥15% of body weight reduction from baseline | Baseline, Week 64 and 84
Percentage of Participants achieving ≥20% of body weight reduction from baseline | Baseline, Week 64 and 84
Change from baseline in Fasting triglycerides | Baseline, Week 64 and 84
Change from baseline in Non-high-density lipoprotein cholesterol (non-HDL-C) | Baseline, Week 64 and 84
Change from baseline in Systolic Blood Pressure (SBP) | Baseline, Week 64 and 84
Change from baseline in Short Form 36 health survey (SF-36) physical function domain score | Baseline, Week 64 and 84
Percent change from baseline in body weight | Baseline, Week 84
Change from baseline in waist circumference | Baseline, Week 64 and 84
Percentage of Participants Achieving HbA1c <7% | Week 64 and Week 84
Percentage of Participants Achieving HbA1c ≤6.5% | Week 64 and Week 84
Percentage of Participants Achieving HbA1c <5.7% | Week 64 and Week 84
Change from Baseline in Fasting Glucose | Baseline, Week 64 and 84
Change from Baseline in Fasting insulin | Baseline, Week 64 and 84
Change from baseline in Total Cholesterol | Baseline, Week 64 and 84
Change from baseline in Low-density lipoprotein cholesterol | Baseline, Week 64 and 84
Change from baseline in Very low-density lipoprotein cholesterol | Baseline, Week 64 and 84
Change from baseline in High-density lipoprotein cholesterol | Baseline, Week 64 and 84
Change from Baseline in Diastolic Blood Pressure (DBP) | Baseline, Week 64 and 84
Percent change from baseline in high-sensitivity C-reactive protein | Baseline, Week 64 and 84
Change from Baseline in EuroQoL 5-Dimension 5-Level (EQ5D-5L) | Baseline, Week 64 and 84
Change from Baseline in Control of Eating Questionnaire (CoEQ) | Baseline, Week 64 and 84
Change from Baseline in Food Noise Questionnaire (FNQ) | Baseline, Week 64 and 84
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Week 84
Number of Participants with Serious adverse events (SAEs) | Week 84
Number of Participants with Adverse Events of Clinical Interest (AECIs) | Week 84
Number of Participants With Clinical Laboratory Abnormalities | Week 84
Number of participants with anti-drug antibodies (ADAs) | Week 84
Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax) of PF-08653944 | Week 84

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests